CLINICAL TRIAL: NCT04375228
Title: An Open-Label, Phase II Multicenter Study of Rituximab or Tocilizumab for Steroid-Dependent Immune-Related Adverse Events Due to Immune Checkpoint Blockade
Brief Title: Study of Rituximab or Tocilizumab for Patients With Steroid-Dependent Immune-Related Adverse Events (irAEs)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Brian Henick, MD, Assistant Professor of Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS9173
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Immune-related Adverse Events; Advanced Solid Tumor
MeSH Terms: interventions — Rituximab; tocilizumab

STUDY DESIGN:
Intervention Model Description: Participants will be assigned either rituximab or tocilizumab based on clinical rationale and consensus recommendation by investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab (Experimental): Patients with histologically confirmed advanced (metastatic or unresectable) solid tumors that have documented irAEs will receive Rituximab.
  Interventions: Drug: Rituximab
- Tocilizumab (Experimental): Patients with histologically confirmed advanced (metastatic or unresectable) solid tumors that have documented irAEs will receive Tocilizumab.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Rituximab — 375mg/m^2 IV weekly for 4 doses
  Other Names: RITUXAN
  Arms: Rituximab
Drug: Tocilizumab — 4mg/kg IV once a month for up to 2 doses
  Other Names: ACTEMRA
  Arms: Tocilizumab

SUMMARY:
The purpose of this study is to examine how effective rituximab or tocilizumab are in treating side effects for people who are receiving immunotherapy treatment requiring prolonged steroid use.

Immune-related side effects are caused by the activation of the immune system. Because rituximab and tocilizumab have been shown to effectively in treating other diseased that involve immune system activation, this study seeks to evaluate how effective they will be in treating immune-related side effects in people receiving immunotherapy treatment for cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and effectiveness of two drugs, either rituximab or tocilizumab, in patients who develop side effects while on treatment with immunotherapy requiring prolonged steroids. Immune-related side effects are caused by activation of the immune system from treatment with immunotherapy. Both rituximab and tocilizumab have been given to patients with autoimmune diseases (diseases where the immune system is activated against normal organs). Immune-related side effects appear to closely mirror these autoimmune conditions.

Participants in this study have developed an immune-related adverse event while on immunotherapy and require a long course of steroids to manage this side effect. Steroids can cause many side effects with prolonged use including problems with sleep, weight gain, diabetes, muscle loss, high blood pressure, high cholesterol, bone loss, and mood disturbances. Drugs such as rituximab and tocilizumab have been shown to be effective in other diseases involving immune system activation. This study is evaluating the effectiveness of these drugs in patients who have immune-related side effects by their ability to help patients discontinue steroids.

ELIGIBILITY:
Inclusion Criteria:

-Patients with histologically confirmed advanced (metastatic or unresectable) solid tumors that develop irAEs secondary to treatment with immune checkpoint inhibitors. Diagnostic evaluation of irAEs must include agreement between medical oncologist and disease-specific subspecialist (e.g. rheumatologist, dermatologist) on therapeutic rationale for either rituximab or tocilizumab-based therapy or if evidence-based indications exist as summarized below: Dermatologic (bullous pemphigoid, pemphigus vulgaris) - Rituximab. Neurologic (autoimmune encephalitis) - Rituximab. Hematologic (immune thrombocytopenia, autoimmune hemolytic anemia) -Rituximab. Rheumatologic (rheumatoid arthritis, psoriatic arthritis) -Rituximab/Tocilizumab.

Renal (autoimmune nephritis) - Rituximab. Pulmonary (pneumonitis) - Tocilizumab. Cardiac (autoimmune myocarditis) - Tocilizumab

-Steroid-dependent, defined as inability to wean less than 10mg of prednisone (or equivalent) after 6 weeks of therapy; patients who develop intolerance to steroids (e.g.

myopathy or hyperglycemia) may be enrolled earlier than 6 weeks at the discretion of the treating physician and/or the principal investigator.

* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Female subject of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use contraception, or abstain from heterosexual activity for the course of the study and through 12 months after last dose of rituximab or 3 months after last dose of tocilizumab. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Males must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 6 months after last dose of rituximab, 180 days even if he has undergone a successful vasectomy
* Vaccinations must be completed 4 weeks prior to the first treatment with rituximab or must not be taken at least 6 months after the last dose of chemotherapy. Non-live vaccines may be given during rituximab treatment; however, patients may experience reduced response rates. The safety of live vaccines has not been studied during cancer treatment and their use is not recommended unless otherwise advised by the oncologist.

Subject must be vaccinated with the pneumococcal vaccine at least 4 weeks prior to initiation of therapy, unless subject was vaccinated within 5 years of study entry. If vaccination occurred greater than 5 years prior to study entry, the subject must be revaccinated at least 4 weeks prior to initiation of therapy

-Have adequate organ and marrow function as defined below: Absolute Neutrophil Count ≥1,000/microliters Platelets ≥100,000 Hemoglobin ≥ 7.0g/dL (without transfusion in past 2 weeks) Note: Patients with cytopenias (e.g immune thrombocytopenia, autoimmune hemolytic anemia) clinically consistent with irAE will be eligible at the discretion of principal investigator. Patients with hematological values below those stated will not receive Tocilizumab aspartate aminotransferase (AST)(SGOT)/ alanine aminotransferase (ALT)(SGPT) ≤2 × institutional upper limit of normal Creatinine clearance of ≥ 30 mL/min. Creatinine clearance (CrCl) should be calculated at screening using the Cockcroft-Gault formula.

Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.

Exclusion Criteria:

* Current participation in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Diagnosis of immunodeficiency or is receiving systemic immunosuppressive therapy other than steroids prior to the first dose of trial treatment
* Treatment with a non-biologic immunosuppressive or immune-modulating drug (e.g. methotrexate, azathioprine, mycophenolate, cyclosporine, hydroxychloroquine, penicillamine) within 4 weeks prior to treatment. Note: Patients who previously received treatment with either rituximab or tocilizumab may receive treatment with the alternative agent after discussion with the treating physician and/or the principal investigator.
* Treatment with other immune-modulating biologic agents within 4 weeks prior to treatment initiation.
* History of anaphylaxis or immunoglobulin E-mediated hypersensitivity to murine proteins or any component of rituximab or tocilizumab History of allergic reactions attributed to compounds of similar chemical or biologic composition to either rituximab or tocilizumab.
* History of human immunodeficiency virus (HIV) infection or other immunodeficiency.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* History of chronic viral hepatitis, alcoholic or metabolic liver disease. Carriers of hepatitis B and patients with a history of hepatitis B infection or positive serology are excluded except in situations where the potential benefit is determined to justify the risk of possible hepatitis B reactivation, which can be fatal. Patients with positive serology should have viral DNA levels checked and a gastrointestinal consultation obtained. If treated with rituximab, such patients should be closely monitored for clinical and laboratory signs of active hepatitis B virus infection and for signs of hepatitis throughout their study participation.
* Central nervous system (CNS) metastases, with the following exception:

Subjects who have previously-treated CNS metastases, are asymptomatic, and have no requirement for steroids in the management of CNS disease (steroids for irAEs are allowed) at least 14 days prior to first dose of study drug. Note: Subjects with carcinomatous meningitis or leptomeningeal spread are excluded regardless of clinical stability.

* History of or current positive purified protein derivative tuberculin skin test (PPD) ( >5mm induration, regardless of Bacille Calmette Guerin (BCG) vaccine administration), or positive QuantiFERON®-TB Gold In-Tube Test (QuantiFERON®), or historical chest x-ray unless completion of treatment has been documented for active tuberculosis (TB), latent TB (a positive test, a negative chest x-ray, and no symptoms or risk factors), unless one month of prophylaxis has been completed prior to inclusion, an indeterminate QuantiFERON® unless followed by a subsequent negative PPD or negative QuantiFERON® as well as a consultation with and clearance by local infectious disease (ID) department
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Transplanted organs (except corneas with transplant performed >3 months prior to screening)
* Active infection, including opportunistic infections, requiring systemic therapy within the past 2 weeks.
* A deep space infection within the past 2 years (including, but not limited to meningitis, epiglottitis, endocarditis, septic arthritis, fasciitis, abdominal or pleural abscess, or osteomyelitis).
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective Institutional Review Board (IRB)approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
* New York Heart Association Classification III or IV heart disease
* Breastfeeding is not permitted during treatment and for 6 months after the last dose of rituximab or 3 months after the last dose of tocilizumab.
* Preexisting central nervous system demyelinating or seizure disorders
* History of diverticulitis, diverticulosis requiring antibiotic treatment, or other symptomatic lower gastrointestinal (GI) conditions that might predispose to perforations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants to Discontinue Steroid Treatment After Rituximab | Up to 8 weeks
  The percentage of participants able to discontinue steroid treatment within 4 weeks after the last dose of Rituximab.
Percentage of Participants to Discontinue Steroid Treatment After Tocilizumab | Up to 12 weeks
  The percentage of participants able to discontinue steroid treatment within 4 weeks after the last dose of Tocilizumab.

SECONDARY OUTCOMES:
Number of Participants with a Change in CTCAE (v5.0) Grade | Up to 24 weeks
  The number of participants with a change in CTCAE (v5.0) grade in participants who develop steroid-dependent immune related adverse events.
The Number Steroid-Dependent Immune-Related Adverse Events | Up to 24 weeks
  To evaluate the safety of rituximab and tocilizumab defined as the number of steroid-dependent immune-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Henick, MD, Principal Investigator — Assistant Professor of Medicine in the Division of Hematology and Oncology
Locations (3):
- United States (3):
  - Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Irving Medical Center, Herbert Irving Comprehensive Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No